CLINICAL TRIAL: NCT06904794
Title: Evaluation of the Gambling Habits of Adolescents and Young Adults Post-COVID-19 and Implementation of a Digital Escape Room Intervention for Preventing Gambling in High School Students: a Mixed-methods Cluster-randomized Controlled Trial (GAMBL-OUT Project)
Brief Title: Evaluation of the Gambling Habits of Adolescents and Young Adults Post-COVID-19 and Implementation of a Digital Escape Room Intervention for Preventing Gambling in High School Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI24/364
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAMBL-OUT escape room (Experimental)
  Interventions: Behavioral: GAMBL-OUT program
- Wait-list control (No Intervention)

INTERVENTIONS:
Behavioral: GAMBL-OUT program — The GAMBL-OUT program consists of two sessions: the first one involves a digital escape room to be delivered in the classroom and a series of physical props to be used during the experience. In small groups (4-5 students), participants need to work together to solve different puzzles and riddles, all of them related to the story of young adults who are dealing with problem gambling. By the end of the game, which will have a limited time (50 minutes), each group will have gained access to a different password. The second session will start from here: each group will share their password so the final puzzle can be solved, and the game will conclude with in a group discussion about what was learned (40 minutes).
  Arms: GAMBL-OUT escape room

SUMMARY:
Gambling behaviors among adolescents and young adults have been experiencing an upward trend in the last years, possibly because of new habits developed during the COVID-19 lockdown restrictions. Different preventive strategies have been proposed: universal classroom-based interventions have shown promising evidence as preventive tools, but challenges exist in engaging the target audience effectively. Serious games, i.e., those designed with the specific intent to educate, broaden knowledge, and change behaviors, have been tested with positive outcomes. Digital escape rooms constitute a modality of serious game that has shown potential for a variety of educational purposes, but their efficacy for preventing addictive behaviors, as well as their long-term impact, has not been widely studied.

The present project aims at assessing the gambling habits of a sample of 16-25-year-olds in the region of Aragon, Spain, that could be compared to the data gathered before the pandemic started, so not only the prevalence rates can be updated but also potential differences in habits (e.g., preferred gambling alternatives) can be detected. This will undoubtedly help the design of effective preventive measures, such as the GAMBL-OUT digital escape room, a serious game to be implemented in high schools with the aim of increasing knowledge, reducing intentions to gamble, and changing attitudes towards gambling.

ELIGIBILITY:
Inclusion Criteria:

* Only high school students aged between 16 and 18
* Being able to read and understand the Spanish language
* Willingness to participate in the study and sign the written informed consent form

Exclusion Criteria:

* Age: <16 years old, or >18 years old

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Problem gambling screening (PGSI) | Baseline
  In the intervention group. This 9-item scale assesses problematic gambling behaviors in the last 12 months and harmful consequences related to gambling. Items are rated on a 4-point scale (0 = never, 3 = almost always). The final score ranges from 0 to 27 and can be interpreted as follows: 0 = non-problem gamblers, 1-2 = low-risk gamblers, 3-7 = moderate-risk gamblers, and 8 and above = problem gamblers).
Problem gambling screening (PGSI) | Three-months follow-up
  In the intervention group. This 9-item scale assesses problematic gambling behaviors in the last 12 months and harmful consequences related to gambling. Items are rated on a 4-point scale (0 = never, 3 = almost always). The final score ranges from 0 to 27 and can be interpreted as follows: 0 = non-problem gamblers, 1-2 = low-risk gamblers, 3-7 = moderate-risk gamblers, and 8 and above = problem gamblers).
Problem gambling screening (PGSI) | Baseline
  In the control group. This 9-item scale assesses problematic gambling behaviors in the last 12 months and harmful consequences related to gambling. Items are rated on a 4-point scale (0 = never, 3 = almost always). The final score ranges from 0 to 27 and can be interpreted as follows: 0 = non-problem gamblers, 1-2 = low-risk gamblers, 3-7 = moderate-risk gamblers, and 8 and above = problem gamblers).
Problem gambling screening (PGSI) | Three-months follow-up
  In the control group. This 9-item scale assesses problematic gambling behaviors in the last 12 months and harmful consequences related to gambling. Items are rated on a 4-point scale (0 = never, 3 = almost always). The final score ranges from 0 to 27 and can be interpreted as follows: 0 = non-problem gamblers, 1-2 = low-risk gamblers, 3-7 = moderate-risk gamblers, and 8 and above = problem gamblers).

SECONDARY OUTCOMES:
Gender | Baseline
  Gender of participants: male, female, other. Both groups
Age | Baseline
  Open-ended question where subjects are asked to indicate numerically their current age. Both groups
Nationality | Baseline
  Country of birth of participants: Spain, other (please specify). Both groups
Current city of residence | Baseline
  Place of current residence: Zaragoza capital, Zaragoza province, Huesca capital, Huesca province, Teruel capita, Teruel province. Both groups
Cohabitation | Baseline
  Who do you live with: first degree relatives (parents, siblings), second degree relatives (grandparents, uncles, aunts, uncles), friends, alone, other (please specify). Both groups
Country of birth of parents | Baseline
  Open-ended question where participants have to indicate in which country their father was born, or where their mother was born. Both groups
Education | Baseline
  Which year of the baccalaureate are you currently in: first or second. Both groups
Employment situation | Baseline
  Indicate how many hours per week you work: no work, between 1 and 10 hours per week, between 11 and 20 hours per week, between 20 and 30 hours per week, between 30 and 40 hours per week. Both groups
Amount of money available for leisure per month | Baseline
  Multiple-choice question ad-hoc where subjects must mark the range of money in euros they have available for leisure. The response options are: 0-100; 101-400; 401-600; 601-1000; 1000 or more. None of the response options is better than the others. In the intervention group
Amount of money available for leisure per month | Baseline
  Multiple-choice question ad-hoc where subjects must mark the range of money in euros they have available for leisure. The response options are: 0-100; 101-400; 401-600; 601-1000; 1000 or more. None of the response options is better than the others. In the control group
Gambling knowledge scale (ad-hoc) | Baseline
  In the intervention group. This questionnaire is composed of 18 separate items that collect information on different aspects of gambling knowledge. Each item is evaluated on a Likert scale with four response options: 'is totally incorrect', 'is incorrect', 'is correct', 'is totally correct'.
Gambling knowledge scale (ad-hoc) | up to 2 weeks
  In the intervention group. This questionnaire is composed of 18 separate items that collect information on different aspects of gambling knowledge. Each item is evaluated on a Likert scale with four response options: 'is totally incorrect', 'is incorrect', 'is correct', 'is totally correct'. There is no overall score on this scale as each item assesses different aspects of gambling knowledge.
Gambling knowledge scale (ad-hoc) | Three-months follow-up
  In the intervention group. This questionnaire is composed of 18 separate items that collect information on different aspects of gambling knowledge. Each item is evaluated on a Likert scale with four response options: 'is totally incorrect', 'is incorrect', 'is correct', 'is totally correct'. There is no overall score on this scale as each item assesses different aspects of gambling knowledge.
Gambling knowledge scale (ad-hoc) | Baseline
  In the control group. This questionnaire is composed of 18 separate items that collect information on different aspects of gambling knowledge. Each item is evaluated on a Likert scale with four response options: 'is totally incorrect', 'is incorrect', 'is correct', 'is totally correct'. There is no overall score on this scale as each item assesses different aspects of gambling knowledge.
Gambling knowledge scale (ad-hoc) | up to 2 weeks
  In the control group. This questionnaire is composed of 18 separate items that collect information on different aspects of gambling knowledge. Each item is evaluated on a Likert scale with four response options: 'is totally incorrect', 'is incorrect', 'is correct', 'is totally correct'. There is no overall score on this scale as each item assesses different aspects of gambling knowledge.
Gambling knowledge scale (ad-hoc) | Three-months follow-up
  In the control group. This questionnaire is composed of 18 separate items that collect information on different aspects of gambling knowledge. Each item is evaluated on a Likert scale with four response options: 'is totally incorrect', 'is incorrect', 'is correct', 'is totally correct'. There is no overall score on this scale as each item assesses different aspects of gambling knowledge.
Ad hoc questions asking attitudes towards gambling | Baseline
  In the intervention group
Ad hoc questions asking attitudes towards gambling | up to 2 weeks
  In the intervention group
Ad hoc questions asking attitudes towards gambling | Three-months follow-up
  In the intervention group
Ad hoc questions asking attitudes towards gambling | Baseline
  In the control group
Ad hoc questions asking attitudes towards gambling | up to 2 weeks
  In the control group
Ad hoc questions asking attitudes towards gambling | Three-months follow-up
  In the control group
Ad hoc questions asking intention to gamble in the future | Baseline
  In the intervention group
Ad hoc questions asking intention to gamble in the future | up to 2 weeks
  In the intervention group
Ad hoc questions asking intention to gamble in the future | Three-months follow-up
  In the intervention group
Ad hoc questions asking intention to gamble in the future | Baseline
  In the control group
Ad hoc questions asking intention to gamble in the future | up to 2 weeks
  In the control group
Ad hoc questions asking intention to gamble in the future | Three-months follow-up
  In the control group
Ad hoc questions asking the gambling habits | Baseline
  In the intervention group
Ad hoc questions asking the gambling habits | Three-months follow-up
  In the intervention group
Ad hoc questions asking the gambling habits | Baseline
  In the control group
Ad hoc questions asking the gambling habits | Three-months follow-up
  In the control group
Implementation outcome: General opinion of the intervention | Three-months follow-up
  The participants indicate their general opinion of the intervention once it is over: 'very positive, I loved it', 'positive, it was a good experience', 'neutral, I was indifferent', 'negative, there were aspects that did not convince me', 'very negative, I was disappointed'. Both groups
Implementation outcome: Ease of use of the platform | Three-months follow-up
  Participants indicate how easy the platform was for them to use: yes or no. Both groups
Implementation outcome: Duration of the intervention | Three-months follow-up
  Opinion on the length of the intervention: 'I thought it was too short', 'I thought it was adequate', 'I thought it was too long'. Both groups
Implementation outcome: Difficulty of the instructions received through the platform | Three-months follow-up
  Opinion on the difficulty of the instructions received through the platform: 'yes', "no", "most yes", "most no". Both groups
Implementation outcome: Amount of information received | Three-months follow-up
  Opinion on the amount of information received: 'excessive', 'adequate', 'insufficient'. Both groups
Implementation outcome: Need for prior knowledge to carry out the intervention | Three-months follow-up
  Opinion on the need for prior knowledge to carry out the intervention: yes or no. Both groups
Implementation outcome: Adequacy of the content of the intervention for the target population | Three-months follow-up
  Opinion on the appropriateness of the content of the intervention for the target population: 'I think it is too easy', 'I think it is suitable for adolescents', 'I think it is too complex', 'other (specify)'. Both groups
Implementation outcome: Effectiveness in conveying information to you about the risks of gambling addiction | Three-months follow-up
  Do you think that the Escape Room has been effective in providing you with information about the risks of gambling addiction?: 'very effective', 'effective', 'neutral', 'not very effective', 'not at all effective'. Both groups
Implementation outcome: Perception of increased knowledge of gambling | Three-months follow-up
  Opinion on perceived increase in knowledge of gambling: 'a lot', 'some', 'a little', 'not at all'. Both groups
Implementation outcome: Integration of educational messages into the dynamics of the Escape Room. | Three-months follow-up
  Opinion on the adequate integration of the educational messages in the Escape Room dynamics: 'quite well', 'well', 'little', 'practically not at all'. Both groups
Implementation outcome: Adequacy of this Escape Room for the prevention of gambling among young people | Three-months follow-up
  Opinion on the suitability of this Escape Room for the prevention of gambling in young people: yes or no. Both groups
Implementation outcome: Opinion on whether participants think it is likely that high schools in Aragon will integrate this Escape Room into their regular programming. | Three-months follow-up
  Opinion on whether participants think it is likely that high schools in Aragon will integrate this Escape Room into their regular programming: yes or no. Both groups
Implementation outcome: Recommendation of this Escape Room to young people in the participants' environment. | Three-months follow-up
  Opinion on whether the participants would recommend this Escape Room to young people in their environment for their training on the functioning and risks of gambling: yes or no. Both groups
Implementation outcome: Consideration of whether this Escape Room is a useful resource for the prevention of gambling among young people. | Three-months follow-up
  Consideration of whether this Escape Room is a useful resource for gambling prevention in young people: yes or no. Both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Spain

REFERENCES:
- [Derived] Barcelo-Soler A, Monreal-Bartolome A, Perez-Aranda A, Campos D, Beltran-Ruiz M, Puebla-Guedea M, Cabrera-Gil I, Garcia-Campayo J, Lopez-Del-Hoyo Y. Evaluation of the gambling habits of Spanish adolescents and young adults post-COVID-19 and implementation of a digital escape room intervention for preventing gambling: study protocol of a cluster-randomized controlled trial (GAMBL-OUT project). BMC Psychol. 2025 Jul 1;13(1):690. doi: 10.1186/s40359-025-03035-x. PMID 40598402